CLINICAL TRIAL: NCT01389635
Title: Abdominoplasty Under Epidural Anesthesia: Safer for the Patient, Easier for the Surgeon.
Brief Title: Abdominoplasty Under Epidural Anesthesia
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Professor Yehuda Ullmann, Head, Department of Plastic Surgery, Rambam Healthcare Campus
Other Study IDs: 0019-11-RMB-CTIL
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Abdominoplasty
Keywords: Abdominoplasty; Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abdominoplasty patients: All patients who underwent abdominoplasty at our institution without concurrent operations

SUMMARY:
Abdominoplasty is one of the most popular body-contouring procedures, yet it is also among the most hazardous aesthetic procedures currently performed. It was shown, in many studies, to be associated with a significant complication rate, some of which are life-threatening. This study describes the investigators experience with a series of abdominoplasties performed under epidural anesthesia. Outcomes are presented, especially in terms of complication, and the practical advantages of this method are discussed.

ELIGIBILITY:
Inclusion Criteria:

* All patients that underwent abdominoplasty between January 2003 and March 2008 in a private hospital by Dr. Yitshak Ramon.

Exclusion Criteria:

* Patients with concurrent operations requiring general anesthesia.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients that underwent abdominoplasty between January 2003 and March 2008 in a private hospital by Dr. Yitshak Ramon.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yitshak Ramon, MD, Principal Investigator — Plastic Surgery Department, Rambam Healthcare Campus
Locations (1):
- Elisha Medical Center, Haifa, Israel